CLINICAL TRIAL: NCT05427136
Title: Prospective Multicentre Cohort Study of Early Pulmonary Dysfunction in Childhood Cancer Patients (SWISS-Pearl Study)
Brief Title: Early Pulmonary Dysfunction in Childhood Cancer Patients
Acronym: SWISS-Pearl
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01206; ks22Usemann
Record Dates: First submitted 2022-06-01; First posted 2022-06-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Dysfunction
Keywords: Childhood cancer; Lung function; Lung imaging; Breath analysis; Exome-wide association studies (EWAS); Genome-wide association studies (GWAS); Pulmotoxic treatment
MeSH Terms: conditions — Neoplasms | interventions — Breath Tests; Magnetic Resonance Imaging; Data Collection; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For study participants who signed further the general consent form, biological materials and health-related data will be coded and stored in a secure biobank/database (BaHOP). The biological material and genetic data are kept in the BaHOP biobank for an indefinite period of time for further, until now not defined research questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung function measurements — All lung function tests are non-invasive and last about 60 minutes per child:
  * Multiple Breath Washout: The nitrogen multiple-breath-washout test (N2MBW) measures ventilation inhomogeneity of the lung that occurs when smaller airways are damaged.
  * Spirometry/Bodyplethysmography/DLCO: Spirometry measures dynamic air flows to quantify airway obstruction of large airways and pulmonary restriction. Plethysmography assesses static lung volumes. Diffusing capacity of the lung for carbon monoxide (DLCO) evaluates diffusion deficits.
Diagnostic Test: Breath Analysis — Patients will exhale into a secondary electrospray-ionization-mass spectrometry (SESI-MS) breath analysis platform. SESI-MS allows real-time breath-printing by detection of both volatile and non-volatile trace components.
Diagnostic Test: Magnetic resonance imaging (MRI) — Functional MRI scan assessing regional fractional lung ventilation and relative perfusion, followed by a morphological MRI scan. This technique allows simultaneous assessment of all affected lung components, the airways, alveoli and pulmonary vasculature.
Other: Standardized interview to assess respiratory symptoms — Short questions on current airway symptoms, recent colds, exercise-related respiratory symptoms, and passive smoking exposure will be assessed. The interview takes about 10 minutes.
Other: Data collection for assessment of clinical parameters and cumulative doses to chemotherapy, radiation, surgery and HSCT — Assessment of clinical parameters and cumulative doses to chemotherapy, radiation, surgery and hematopoietic stem cell transplantation (HSCT). Data on cumulative doses of pulmotoxic chemotherapy (carmustine, lomustine, busulfan, bleomycin, methotrexate and cyclophosphamide, fludarabine, ifosfamide, melphalan and thiotepa) and radiation therapy at the region of the chest from patient's hospital charts will be collected. Information on chest wall and lung surgery will be retrieved from the surgical reports. Information about conditioning regimens including cumulative chemotherapy doses and total body irradiation of patients undergoing HSCT will be collected. Further information on the health state of the patient and interventions (e.g. development of pneumonia, antibiotic treatment) will be collected from the hospital charts.
Other: Collection of genetic samples — Germline DNA is collected (e.g. through saliva or buccal cell sampling) for later analysis on genetic risk factors for pulmonary complications.

SUMMARY:
This longitudinal, prospective, multicentre study is to monitor lung function prospectively in childhood cancer patients after diagnosis. The impact of cancer treatment on pulmonary dysfunction non-invasively using lung function, lung imaging and breath analysis as well as clinical symptoms using a questionnaire will be assessed at different time points.

ELIGIBILITY:
Inclusion Criteria:

* at least one of the following cancer treatments:

  * chest radiation
  * treatment with any kind of chemotherapy
  * hematopoietic stem cell transplantation (HSCT)
  * thoracic surgery
* consent for Childhood Cancer Registry (ChCR) registration

Exclusion Criteria:

* no signed informed consent
* Operation outside the chest area as only cancer treatment
* Relapsed cancer (patients who develop relapse during the study will not be excluded)
* In addition for MRI and lung function tests:

  * Subjects who are respiratory insufficient and cannot perform a lung function test (less than 92% O2 saturation; under O2 therapy)
  * Pregnant
  * MRI measurement not possible without sedation
  * Metal (e.g. pacemaker) in the body

Ages: 4 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Every new diagnosed cancer patient and every cancer patient planned for HSCT who is 4 years or older will be asked by the paediatric oncologist to participate in the study. This study will be conducted at the University Children's Hospital of Basel, Bern, Geneva, Lausanne and Zürich.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2051-06 (Estimated); Study Completion 2051-06 (Estimated)

PRIMARY OUTCOMES:
Change in Forced expiratory volume in 1 second (FEV1) | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Dynamic lung function parameter: Forced expiratory volume in 1 second (FEV1)
Change in ratio of FEV1/forced vital capacity (FVC) for airway obstruction | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Dynamic lung function parameter: ratio of FEV1/forced vital capacity (FVC) for airway obstruction
Change in total lung capacity (TLC) | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Static lung function parameter: total lung capacity (TLC) to assess lung restriction
Change in residual volume (RV)/TLC | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Static lung function parameter: residual volume (RV)/TLC to assess hyperinflation
Change in lung clearance index (LCI) | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Global ventilation inhomogeneity assessed by lung clearance index (LCI)
Change in Alveolar-capillary membrane diffusion | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Alveolar-capillary membrane diffusion
Change in percentage portion of the lung volume with impaired ventilation or perfusion | Before start of therapy, 12 months after end of intensive treatment,24 months after end of intensive treatment
  Functional MRI: the primary outcome of functional lung imaging is the percentage portion of the lung volume with impaired ventilation or perfusion.
Change in lung morphology assessed by MRI | Before start of therapy, 12 months after end of intensive treatment,24 months after end of intensive treatment
  Change in lung morphology assessed by MRI (description of structural changes: ground glass changes, thickened septal lines, interstitial infiltrates, diffuse alveolar infiltrates, haemorrhage, focal consolidation, fibrosis, pulmonary hypertension, pleural effusion, nodular changes, vasculitis (wall thickening) and thrombosis will be assessed)

SECONDARY OUTCOMES:
Change in 4-hydroxy-2-nonenal in exhaled breath | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Breath analysis: 4-hydroxy-2-nonenal is regarded as a surrogate marker for oxidative stress in the human body.
Change in volatile organic compounds (VOCs) in exhaled breath | At Baseline (start of therapy), at month 3 (during intensive treatment), at month 6-18 (end of intensive treatment), 12 months after end of intensive treatment,24 months after end of intensive treatment
  Untargeted explorative approach to assess volatile organic compounds (VOCs) in exhaled breath
Assessment of genetic variants through saliva or buccal cell sampling (collection of germline DNA) | At Baseline (start of therapy)
  Genetic variants associated with susceptibility to cancer therapy or related to lung development. Assessed in the Germline DNA Biobank Switzerland for childhood cancer and blood disorders (BISKIDS, as part of the Paediatric Biobank for Research in Haematology and Oncology [BaHOP], ethics approval PB_2017-00533 to assess genetic determinants of pulmonary toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Usemann, PD Dr. med., Principal Investigator — University Children's Hospital Basel, UKBB
Locations (5):
- Switzerland (5):
  - University Children's Hospital Basel (UKBB), Basel
  - Universitätsklinik für Kinderheilkunde, Bern
  - Geneva University Hospital, Geneva
  - Centre hospitalier universitaire vaudois Lausanne, Lausanne
  - Universitäts-Kinderspital Zürich, Zurich